CLINICAL TRIAL: NCT05851534
Title: Preoperative Optimisation of Modifiable Risk Factors in Surgery of the Pancreas: the Implementation of Best Practice Before Pancreatic Resection
Brief Title: Preoperative Optimisation of Modifiable Risk Factors in Surgery of the Pancreas
Acronym: PROMISE-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Rising Tide Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2023-3607
Record Dates: First submitted 2023-04-14; First posted 2023-05-09 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Prehabilitation; Pancreas Cancer; Surgery; Postoperative Complications
Keywords: Prehabilitation; Pancreas; Preoperative optimisation
MeSH Terms: conditions — Pancreatic Neoplasms; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized superiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care (No Intervention): Receiving standard preoperative care
- Best practice program (Experimental): Implementation of best practice preoperative optimisation program
  Interventions: Behavioral: Preoperative optimisation program

INTERVENTIONS:
Behavioral: Preoperative optimisation program — Preoperative screening of all patients scheduled for pancreatic resection on (aerobic) fitness level, malnutrition risk, psychological resilience, haemoglobin, iron and HbA1c concentration, frailty, and alcohol and smoking behaviour. All patients are provided with a patient-tailored, multimodal prehabilitation program, in which these potentially (partly) modifiable factors are preoperatively addressed
  Arms: Best practice program

SUMMARY:
The goal of this stepped-wedge randomized controlled trial is to investigate whether implementation of a best practice program for preoperative optimisation (prehabilitation program) with a focus on screening, assessment, and intervention of 8 potentially (partly) modifiable risk factors in patients with (suspected) pancreatic cancer will improve outcome. The main questions it will aim to answer are:

1. Does a prehabilitation program improve the time to functional recovery after pancreatic surgery?
2. Does a prehabilitation program lead to a reduction in the Comprehensive Complication Index after pancreatic surgery?

DETAILED DESCRIPTION:
Background In the past, little attention has been given in the daily practice to the patient's condition before an operation. Recent studies have shown the benefit of preoperative optimisation programs. However, these studies consisted only of smaller studies and were mainly performed in patients who underwent colorectal surgery. Although promising, unfortunately, strong evidence to support the contribution of prehabilitation to optimize the functional outcome after surgery is still lacking and consequently it is not included in the Dutch basic health insurance package.

Objective To investigate whether implementation of a best practice program for preoperative optimisation of patients with a focus on screening, assessment, and intervention of 8 potentially (partly) modifiable risk factors (low (aerobic) fitness level, malnutrition, low psychological resilience, comorbidities (iron deficiency (anaemia), impaired glucose control and frailty), and intoxications (alcohol and smoking behaviour)) will improve the time to functional recovery.

Study design A nationwide stepped-wedge cluster randomized trial. In this design all participating centres will cross over from current practice to the best practice program, in a randomised order. At the end of the study, all centres will have implemented the best practice program.

Study population 13 centres performing major pancreatic surgery in the Netherlands collaborating within the Dutch Pancreatic Cancer Group (DPCG).

Intervention Preoperative screening of all patients scheduled for pancreatic resection on (aerobic) fitness level, malnutrition risk, psychological resilience, haemoglobin, iron and HbA1c concentration, frailty, and alcohol and smoking behaviour. All patients are provided with a patient-tailored, multimodal prehabilitation program, in which these potentially (partly) modifiable factors are preoperatively addressed. This program is based on findings in previous screening and prehabilitation programs, a national inventory of current preoperative care protocols and expert opinion. Consensus upon this program was reached with pancreatic surgeons from all centres of the DPCG. The final program was critically reviewed by the advisory committee of internationally respected experts in the field of prehabilitation and pancreatology.

Comparison Preoperative care according to current practice.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are planned for a curative treatment with or without neoadjuvant treatment and elective pancreatic resection in one of the centres of the Dutch Pancreatic Cancer Group (i.e. all centres performing major pancreatic surgery)

Exclusion Criteria:

* age < 18 years
* acute pancreatic resections (resection scheduled within two weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2575 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2027-09-02 (Estimated); Study Completion 2028-09-02 (Estimated)

PRIMARY OUTCOMES:
Time to functional recovery | On average 6-10 days
  Functional recovery is achieved when all of the following five criteria are met:
  a) restored level of mobility at the preoperative level, b) sufficient pain control with oral medication alone, c) ability to maintain at least 50% daily required energy intake, d) no intravenous fluid administration, and e) no clinical signs of infection.

SECONDARY OUTCOMES:
Comprehensive Complication Index (CCI) | 30 days postoperative
  The CCI is calculated as the sum of all complications that are weighted for their severity, with a range from 0 to 100, whereby a higher score indicates presence of more complications and/or more severe complications.
Length of hospital stay | On average 2 weeks postoperative
  Length of hospital stay of the primary admission, measured in days
Readmissions | 30 days after discharge of primary admission
  Readmissions within 30 days after discharge
Postoperative complications | During primary admission, on average 14 weeks postoperative
  Any postoperative complication
Incremental cost-effectiveness ratio (ICER) | 1 year postoperative
  The difference in costs between standard care and best practice care divided by the difference in health benefits, measured in quality-adjusted life years (QALYs).
Evaluation of health status | At baseline, 3 months and 12 months postoperative
  Reported health status measured with questionnaire EQ-5D-5L
Evaluation of quality of life for cancer patients | At baseline, 3 months and 12 months postoperative
  Reported quality of life measured with questionnaire EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Marcel den Dulk, MD PhD, Principal Investigator — Maastricht University Medical Center/ University Maastricht
Locations (13):
- Netherlands (13):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Amsterdam University Medical Center, Amsterdam
  - OLVG, Amsterdam
  - Amphia Hospital, Breda
  - Catharina Hospital, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leiden University Medical Center, Leiden
  - Maatricht University Medical Center, Maastricht
  - Radboud University Medical Center, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - RAKU, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be shared, after deidentification upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Data will be available upon request. Request should be directed to marcel.den.dulk@mumc.nl.